CLINICAL TRIAL: NCT05553184
Title: Activation of Brown Adipose Tissue Thermogenesis in Humans Using Formoterol Fumarate, a Beta-2 Adrenergic Receptor Agonist
Brief Title: Activation of Brown Adipose Tissue Thermogenesis in Humans Using Formoterol Fumarate (GB10)
Acronym: GB10
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, André Carpentier, Tenure professor, Université de Sherbrooke
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: GB10-2021-3873
Record Dates: First submitted 2022-08-25; First posted 2022-09-23 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Brown adipose tissue; formoterol fumarate; Thermogenesis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Niacin; Tablets; Positron-Emission Tomography; Absorptiometry, Photon; Biopsy

STUDY DESIGN:
Intervention Model Description: The protocol will be carried out as a within-subject, randomized, cross-over study in which each subject will serve as his/her own control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acute Cold Exposure (Active Comparator): 3h-acute cold exposure.
  Interventions: Other: Acute Cold Exposure; Diagnostic Test: Positron Emission Tomography (PET); Diagnostic Test: Indirect calorimetry; Diagnostic Test: dual-energy x-ray absorptiometry (DEXA scan); Procedure: Biopsy; Procedure: iv lines; Procedure: Electromyogram (EMG)
- Formoterol with nicotinic acid (Experimental): Formoterol fumarate or Oxeze® Turbuhaler®: 48 µg (4 inhalations of 12 µg).
  Nicotinic acid or Niacin: repeated doses of 150 MG every 30 minutes, for 3 hours.
  Interventions: Drug: Formoterol Fumarate 12 micrograms Inhalation Powder; Drug: Nicotinic Acid 50 MG Oral Tablet; Diagnostic Test: Positron Emission Tomography (PET); Diagnostic Test: Indirect calorimetry; Procedure: Biopsy; Procedure: iv lines
- Formoterol without nicotinic acid (Experimental): Formoterol fumarate or Oxeze® Turbuhaler®: 48 µg (4 inhalations of 12 µg).
  Interventions: Drug: Formoterol Fumarate 12 micrograms Inhalation Powder; Diagnostic Test: Positron Emission Tomography (PET); Diagnostic Test: Indirect calorimetry; Procedure: Biopsy; Procedure: iv lines

INTERVENTIONS:
Drug: Formoterol Fumarate 12 micrograms Inhalation Powder — At time 60 minutes, a total of 48 micrograms will be inhaled within 3 minutes: 4 inhalations of 12 micrograms of fumarate formoterol (Oxeze® Turbuhaler®).
  Other Names: Oxeze Turbuhaler
  Arms: Formoterol with nicotinic acid; Formoterol without nicotinic acid
Drug: Nicotinic Acid 50 MG Oral Tablet — a total dose of 1050 MG will be ingested. From time 0 to 180 minutes, doses of 150 MG will be repeated every 30 minutes.
  Other Names: Niacin 50 MG
  Arms: Formoterol with nicotinic acid
Other: Acute Cold Exposure — Participants will be fitted with a liquid-conditioned tube suit. The liquid-conditioned tube suit will be perfused with 18°C water using a temperature- and flow-controlled circulation bath from time 0 to 180 min.
  Arms: Acute Cold Exposure
Diagnostic Test: Positron Emission Tomography (PET) — PET imaging using C11-palmitate (time 90), C11-acetate (time 120) and F18-Fluorodeoxyglucose (FDG) (time 150)
Diagnostic Test: Indirect calorimetry — will be repeated every hour, for 20 minutes, using Vmax29n.
Diagnostic Test: dual-energy x-ray absorptiometry (DEXA scan) — Whole body scan
  Arms: Acute Cold Exposure
Procedure: Biopsy — After local anesthesia with 2% xylocaine without epinephrine, 100-200 mg of subcutaneous adipose tissue will be sampled by needle (14G) biopsy
Procedure: iv lines — for stable tracer perfusion and blood sampling
Procedure: Electromyogram (EMG) — Surface electrodes will be used to measure skeletal muscle activity and shivering intensity
  Arms: Acute Cold Exposure

SUMMARY:
One emerging, highly modifiable homeostatic mechanism for energy expenditure in humans is brown adipose tissue (BAT) thermogenesis. BAT is currently considered a prime target for the treatment of obesity and Type 2 diabetes (T2D).

Using acetate and fluorodeoxyglucose (FDG) positron emission tomography (PET) , It has been demonstrated that BAT thermogenesis is inducible by chronic cold exposure.

BAT activation through cold exposure is associated with improved glucose homeostasis and insulin sensitivity.

A pharmaceutical approach, which seemed to be very promising to stimulate the activation of BAT, was the use of a selective beta 3-adrenergic receptor agonist, mirabegron. Nevertheless, in a later study, It has been demonstrated that human BAT thermogenesis is under the control of beta-2, not beta-3, adrenergic receptor. The most selective beta-2 adrenergic receptor agonist approved for clinical use in Canada is formoterol fumarate, given in inhalation for the treatment of asthma (Oxeze®).

In summary, BAT contributes to cold-induced thermogenesis and is recruited by chronic cold exposure as well as by a growing number of food supplements and drugs. Intracellular triglyceride (TG) is the primary source of fuel for BAT thermogenesis under normal physiological conditions, as blocking intracellular TG lipolysis using nicotinic acid abolishes BAT thermogenesis. Beta-2 adrenergic stimulation is the pharmacological target to activate BAT thermogenesis in humans and may also lead to white adipose tissue lipolysis. Using a highly-selective beta-2 receptor agonist with and without administration of nicotinic acid would thus give the opportunity to quantify more precisely energy expenditure accounted by BAT thermogenesis and white adipose tissue metabolism in humans.

DETAILED DESCRIPTION:
Each participant will undergo three metabolic sessions with PET imaging using [11C]-palmitate, [11C]-acetate and [18F]-FDG:

1. during a 3-h cold exposure (Study A, control condition)
2. after inhalation of Formoterol with oral nicotinic acid (Study B)
3. after inhalation of Formoterol only (Study C).

ELIGIBILITY:
Inclusion Criteria:

* BMI of 18 to 30 kg/m2.

Exclusion Criteria:

* Change in weight of more than 2 kg over the past 3 months or recent changes in lifestyle;
* The presence of any chronic medical condition requiring any pharmacological treatment;
* Previous intolerance or allergy to lactose, formoterol, nicotinic acid or local anesthetic agent;
* Any previous cardiac arrhythmia, long QT syndrome or hypokalemia;
* Chronic treatment with any medication other than contraceptives;
* Acute use of any drug other that acetaminophen or non-steroidal anti-inflammatory without decongestant or other stimulants;
* Smoking or consumption of more than 2 alcoholic beverages per day;
* Having participated to a research study with exposure to radiation in the last two years before the start of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
Change in Brown Adipose Tissue thermogenesis (formoterol induced, cold-induced and effect of nicotinic acid) | measured 60 minutes before and 90 minutes after cold exposure (A) and 30 minutes after inhalation of Fumarate Formoterol (B and C)
  determined using [11C]-acetate PET

SECONDARY OUTCOMES:
Brown Adipose Tissue (BAT) glucose uptake | measured 150 minutes after the start of acute cold exposure (A), and 90 minutes after inhalation of Fumarate Formoterol (B and C)
  determined using [18F]-FDG dynamic PET acquisition
Brown Adipose Tissue nonesterified fatty acid (NEFA) metabolism (uptake, oxidation, esterification and release rates) | measured 120 minutes after the start of acute cold exposure (A), and 60 minutes after inhalation of Fumarate Formoterol (B and C)
  determined using [11C]-palmitate PET method
Change in systemic plasma NEFA turnover. | measured at baseline and every 60 minutes after the start of acute cold exposure (A) and every 60 minutes after inhalation of fumarate formoterol (B and C), for 4 hours
  Determined using continuous infusion of labelled palmitate from time -60 to 180.
Change in systemic plasma glycerol turnover. | measured at baseline and every hour after the start of acute cold exposure (A) and every hour after inhalation of fumarate formoterol (B and C), for 4 hours.
  Determined using continuous infusion of [1,1,2,3,3-D2]-glycerol from time -60 to 180 .
Change in systemic plasma glucose turnover. | measured at baseline and every hour after the start of acute cold exposure (A) and every hour after inhalation of fumarate formoterol (B and C), for 5.50 hours
  Determined using continuous infusion of [6,6 D2]-glucose from time -150 to 180 .
BAT triglyceride content | measured 180 minutes after the start of cold exposure (A) and 90 minutes after inhalation of fumarate formoterol (B and C)
  Determined using the CT radio-density method
Change in whole-body energy expenditure | measured at baseline and every hour after the start of acute cold exposure (A) and every hour after inhalation of fumarate formoterol (B and C), for 4 hours
  Determined using indirect calorimetry
Muscle shivering activity | measured at baseline and every hour after the start of acute cold exposure (A) and every hour after inhalation of fumarate formoterol (B and C), for 4 hours
  Determined using the surface electromyogram (EMG)
Change in insulin sensitivity | measured at baseline and every 60 minutes after the start of acute cold exposure (A) and every 60 minutes after inhalation of fumarate formoterol (B and C), for 4 hours.
  Determined by measuring circulating glucose, NEFA, insulin and C-peptide
Protein expression of subcutaneous abdominal white adipose tissue | measured at baseline and 180 minutes after the start of the cold exposure (study A) and 120 minutes after inhalation of fumarate formoterol (study B and C)
  Using biopsy

CONTACTS AND LOCATIONS:
Overall Officials: André C. Carpentier, M.D., Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche du CHUS, Sherbrooke, Quebec, Canada